CLINICAL TRIAL: NCT05927662
Title: Does the Sagittal Profile of the Patient Effect the Results of Mini-open Lumbar Discectomy? A Preliminary Mid-term Results Report
Brief Title: Results of Mini-open Discectomy According to Sagittal Profile
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İsmail Demirkale, clinical professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2012KAEK15-2603
Record Dates: First submitted 2023-06-08; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Displacement of Intervertebral Disc Without Myelopathy
Keywords: intervertebral disc displacement, spinal curvatures, Outcome
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Curvatures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2: Patients with Roussouly type 2 sagittal profile
  Interventions: Procedure: lumbar discectomy
- Type 1,3,4: Patients with other Roussouly type sagittal profiles (1,3,4)
  Interventions: Procedure: lumbar discectomy

INTERVENTIONS:
Procedure: lumbar discectomy — mini-open discectomy

SUMMARY:
In the normal healthy population, the sagittal alignment can be divided into four types based on the size of the sacral slope and lumbar lordosis. The effect of this sagittal profile especially type 2 with almost straight lordosis on the clinical outcomes of patients after mini-open discectomy is unknown. In this study, the results of patients who underwent mini-open discectomy were evaluated according to sagittal profile types of the patients.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is the most common cause of sciatica and when conservative treatment fails or there is progressive neurological deficit, surgical excision of the herniated nucleosus pulposus is standard of care. Although minimally invasive methods such as endoscopic discectomy have been tried to be popular in recent years, open lumbar discectomy is still successfully performed in lumbar disc herniations due to some drawbacks of endoscopic techniques such as having long learning curve, higher radiation exposure to the surgeon, similar long-term results or the deception of commercial enterprises about endoscopic techniques and the pressure placed on surgeons in this direction.

Herniation of the nucleus pulposus as a result of massive LDH will inevitably result in disruption of normal lumbar biomechanics. Moreover, it has been shown that the healing process of the posterolateral herniation, which is biologically the weakest part of the posterior longitudinal ligament, will cause disc degeneration as a result of the repair and inflammation process in the annulus. However, the same authors claimed that, unlike the process in discogenic low back pain, macrophages in herniated discs can act to remove free pulposus fragments. There are few studies in the literature about the long-term consequences of this degeneration, which the investigators can consider as an accelerated aging process. Although clinically very successful results are obtained in the early postoperative period, it has been reported that the long-term success after discectomy may decrease from 90% to 60% over time. Depression or somatization, strenuous job and recurrent disc herniation or degeneration have been shown to cause long-term regression of results. In a prospective cohort study the authors reported a similar or worse leg pain rate in 30% of patients at the end of 10 years. In a study investigating reoperation after open lumbar discectomy, it was reported that the estimated rate of reoperation reached almost 45% at the end of 30 years.

In an extraordinary review evaluating the spinopelvic organization and the pathological adaptation to it, the mechanical stress, especially increased by hypolordosis, would cause the degenerative process in the spine to progress more rapidly. The basic theories explaining this are that the contact force, which is defined as the resultant force of the system created by gravity and abdominal pressure from the front and the dense paraspinal muscle mass from the posterior, mainly targets the discs. However, studies evaluating spinopelvic orientation in patients with LDH are limited. In a case-control study investigating the relationship between sciatica and spinopelvic harmony, more vertical sacrum, anterior C7 plumb line and hypolordosis were found in the LDH group. In a study examining the etiology and mechanism of sagittal imbalance caused by LDH, lumbar lordosis improved almost twice after endoscopic discectomy and LDH is probably one of the causes of compensatory sagittal imbalance.

Although there are studies on the pathogenesis and mechanics of LDH's etiology and post-discectomy results, the effect of the generally accepted normal lordosis types described by Roussouly P. on the degenerative process and patient scores after open standard discectomy is unknown. Therefore, in this study, the investigators aimed to compare the clinical results of patients with hypolordotic Type 2 and other types after open discectomy. Our hypothesis is that the mid-term clinical scores will be worse in Roussouly Type 2 patients with less lordosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete skeletal maturation (>18 years)
* Lumbar disc herniation with >50% canal narrowing
* Severe leg and back pain associated with large LDH
* >6 weeks of unsuccessful conservative treatment
* Signed a written consent form

Exclusion Criteria:

* Patients with spondyloarthropathy
* Recurrent disc herniation
* Spinal instability
* >10 degrees of coronal deformity
* Incomplete data in the records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with lumbar disc herniation who are candidates for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | change between preoperative and postoperative last (12th month) control
  quantify disability for low back pain
Japanese Orthopedic Association scores | at 12th month control
  a simple scoring measure for radiculopathy with 29 points: Excellent neurological function 25-28 points: Good neurological function 17-24 points: Fair neurological function 11-16 points: Poor neurological function 10 points and below: Bad neurological function

SECONDARY OUTCOMES:
Body mass index (kg/cm2) | preoperative
  demographic characteristic
abdominal diameter | preoperative
  radiological assessment of coronal abdominal diameter, cm
classification of disc degeneration | change between preoperative and at 12th month control
  Pfirrmann grading scale for intervertebral disc degeneration where Grade I: Normal disc appearance with high signal intensity, a smooth contour, and high water content.
  Grade II: Mild signs of degeneration with slightly decreased high signal intensity compared to normal discs.
  Grade III: Moderate degeneration with an irregular contour, further decreased high signal intensity, and possible small fissures within the disc.
  Grade IV: Severe degeneration with a more pronounced irregularity, significant decrease in high signal intensity, and presence of larger fissures and herniations within the disc.
  Grade V: Advanced degeneration with a substantially decreased signal intensity, loss of contour, and structural integrity of the disc. Large herniations may be present within the disc.
visual analogue scale | change between preoperative and postoperative 1st, 6th and 12th month controls
  pain rating scale from 0 (no pain) to 10 (maximum pain)
Tanita-SC 240 body analysis | preoperative and 12th month control
  Body fat percentages of the patients
sagittal abdominal diameter | preoperatively
  radiological assessment of sagittal abdominal diameter, cm
ventral subcutaneous thickness | preoperatively
  radiological assessment of ventral fat thickness, cm
Adjacent muscle cross-sectional areas (cm2) | preoperatively
  Musculus Multifidus, Erector spina and Psoas muscle cross-sectional areas

CONTACTS AND LOCATIONS:
Overall Officials: süheyla atay, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Atatürk Sanatoryum SUAM, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gadjradj PS, Harhangi BS, Amelink J, van Susante J, Kamper S, van Tulder M, Peul WC, Vleggeert-Lankamp C, Rubinstein SM. Percutaneous Transforaminal Endoscopic Discectomy Versus Open Microdiscectomy for Lumbar Disc Herniation: A Systematic Review and Meta-analysis. Spine (Phila Pa 1976). 2021 Apr 15;46(8):538-549. doi: 10.1097/BRS.0000000000003843. PMID 33290374
- [Result] Ropper AH, Zafonte RD. Sciatica. N Engl J Med. 2015 Mar 26;372(13):1240-8. doi: 10.1056/NEJMra1410151. No abstract available. PMID 25806916
- [Result] Hsu HT, Chang SJ, Yang SS, Chai CL. Learning curve of full-endoscopic lumbar discectomy. Eur Spine J. 2013 Apr;22(4):727-33. doi: 10.1007/s00586-012-2540-4. Epub 2012 Oct 17. PMID 23076645
- [Result] Ahn Y, Kim CH, Lee JH, Lee SH, Kim JS. Radiation exposure to the surgeon during percutaneous endoscopic lumbar discectomy: a prospective study. Spine (Phila Pa 1976). 2013 Apr 1;38(7):617-25. doi: 10.1097/BRS.0b013e318275ca58. PMID 23026867
- [Result] Gadjradj PS, Rubinstein SM, Peul WC, Depauw PR, Vleggeert-Lankamp CL, Seiger A, van Susante JL, de Boer MR, van Tulder MW, Harhangi BS. Full endoscopic versus open discectomy for sciatica: randomised controlled non-inferiority trial. BMJ. 2022 Feb 21;376:e065846. doi: 10.1136/bmj-2021-065846. PMID 35190388
- [Result] Peng B, Hao J, Hou S, Wu W, Jiang D, Fu X, Yang Y. Possible pathogenesis of painful intervertebral disc degeneration. Spine (Phila Pa 1976). 2006 Mar 1;31(5):560-6. doi: 10.1097/01.brs.0000201324.45537.46. PMID 16508552
- [Result] Benzakour A, Benzakour T. Lumbar disc herniation: long-term outcomes after mini-open discectomy. Int Orthop. 2019 Apr;43(4):869-874. doi: 10.1007/s00264-019-04312-2. Epub 2019 Mar 8. PMID 30848331
- [Result] Prolo DJ, Oklund SA, Butcher M. Toward uniformity in evaluating results of lumbar spine operations. A paradigm applied to posterior lumbar interbody fusions. Spine (Phila Pa 1976). 1986 Jul-Aug;11(6):601-6. doi: 10.1097/00007632-198607000-00012. PMID 3787326
- [Result] Guo JJ, Yang H, Tang T. Long-term outcomes of the revision open lumbar discectomy by fenestration: A follow-up study of more than 10 years. Int Orthop. 2009 Oct;33(5):1341-5. doi: 10.1007/s00264-008-0648-2. Epub 2008 Oct 14. PMID 18853159
- [Result] Loupasis GA, Stamos K, Katonis PG, Sapkas G, Korres DS, Hartofilakidis G. Seven- to 20-year outcome of lumbar discectomy. Spine (Phila Pa 1976). 1999 Nov 15;24(22):2313-7. doi: 10.1097/00007632-199911150-00005. PMID 10586454
- [Result] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of sciatica secondary to a lumbar disc herniation: 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):927-35. doi: 10.1097/01.brs.0000158954.68522.2a. PMID 15834338
- [Result] Son IN, Kim YH, Ha KY. Long-term clinical outcomes and radiological findings and their correlation with each other after standard open discectomy for lumbar disc herniation. J Neurosurg Spine. 2015 Feb;22(2):179-84. doi: 10.3171/2014.10.SPINE131126. Epub 2014 Nov 28. PMID 25431963
- [Result] Roussouly P, Pinheiro-Franco JL. Biomechanical analysis of the spino-pelvic organization and adaptation in pathology. Eur Spine J. 2011 Sep;20 Suppl 5(Suppl 5):609-18. doi: 10.1007/s00586-011-1928-x. Epub 2011 Aug 2. PMID 21809016
- [Result] Endo K, Suzuki H, Tanaka H, Kang Y, Yamamoto K. Sagittal spinal alignment in patients with lumbar disc herniation. Eur Spine J. 2010 Mar;19(3):435-8. doi: 10.1007/s00586-009-1240-1. Epub 2009 Dec 20. PMID 20091188
- [Result] Liang C, Sun J, Cui X, Jiang Z, Zhang W, Li T. Spinal sagittal imbalance in patients with lumbar disc herniation: its spinopelvic characteristics, strength changes of the spinal musculature and natural history after lumbar discectomy. BMC Musculoskelet Disord. 2016 Jul 22;17:305. doi: 10.1186/s12891-016-1164-y. PMID 27444272
- [Result] Roussouly P, Gollogly S, Berthonnaud E, Dimnet J. Classification of the normal variation in the sagittal alignment of the human lumbar spine and pelvis in the standing position. Spine (Phila Pa 1976). 2005 Feb 1;30(3):346-53. doi: 10.1097/01.brs.0000152379.54463.65. PMID 15682018
- [Result] Pfirrmann CW, Metzdorf A, Zanetti M, Hodler J, Boos N. Magnetic resonance classification of lumbar intervertebral disc degeneration. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1873-8. doi: 10.1097/00007632-200109010-00011. PMID 11568697
- [Result] van den Hout WB, Peul WC, Koes BW, Brand R, Kievit J, Thomeer RT; Leiden-The Hague Spine Intervention Prognostic Study Group. Prolonged conservative care versus early surgery in patients with sciatica from lumbar disc herniation: cost utility analysis alongside a randomised controlled trial. BMJ. 2008 Jun 14;336(7657):1351-4. doi: 10.1136/bmj.39583.709074.BE. Epub 2008 May 23. PMID 18502912
- [Result] Berthonnaud E, Dimnet J, Roussouly P, Labelle H. Analysis of the sagittal balance of the spine and pelvis using shape and orientation parameters. J Spinal Disord Tech. 2005 Feb;18(1):40-7. doi: 10.1097/01.bsd.0000117542.88865.77. PMID 15687851
- [Result] Laouissat F, Sebaaly A, Gehrchen M, Roussouly P. Classification of normal sagittal spine alignment: refounding the Roussouly classification. Eur Spine J. 2018 Aug;27(8):2002-2011. doi: 10.1007/s00586-017-5111-x. Epub 2017 Apr 28. PMID 28455623
- [Result] Pizones J, Martin MB, Perez-Grueso FJS, Yilgor C, Vila-Casademunt A, Serra-Burriel M, Obeid I, Alanay A, Acaroglu ER, Pellise F; ESSG European Spine Study Group. Impact of Adult Scoliosis on Roussouly Sagittal Shape Classification. Spine (Phila Pa 1976). 2019 Feb 15;44(4):270-279. doi: 10.1097/BRS.0000000000002800. PMID 30020277
- [Result] Wu J, Chen Z, Wang H, Tian Y, Ma X, Lyu F, Jiang J, Wang H. The Influence of Roussouly Type on the Prevalence, Subtype, and Distribution Characteristics of Modic Changes in Patients with Lumbar Degenerative Disc Disease. World Neurosurg. 2023 Jan;169:e102-e109. doi: 10.1016/j.wneu.2022.10.070. Epub 2022 Oct 26. PMID 36309336
- [Result] Zhang F, Zhang K, Tian HJ, Wu AM, Cheng XF, Zhou TJ, Zhao J. Correlation between lumbar intervertebral disc height and lumbar spine sagittal alignment among asymptomatic Asian young adults. J Orthop Surg Res. 2018 Feb 12;13(1):34. doi: 10.1186/s13018-018-0737-x. PMID 29433530
- [Result] Amin RM, Andrade NS, Neuman BJ. Lumbar Disc Herniation. Curr Rev Musculoskelet Med. 2017 Dec;10(4):507-516. doi: 10.1007/s12178-017-9441-4. PMID 28980275
- [Result] Takatalo J, Karppinen J, Taimela S, Niinimaki J, Laitinen J, Sequeiros RB, Samartzis D, Korpelainen R, Nayha S, Remes J, Tervonen O. Association of abdominal obesity with lumbar disc degeneration--a magnetic resonance imaging study. PLoS One. 2013;8(2):e56244. doi: 10.1371/journal.pone.0056244. Epub 2013 Feb 13. PMID 23418543
- [Result] Warnberg J, Nova E, Moreno LA, Romeo J, Mesana MI, Ruiz JR, Ortega FB, Sjostrom M, Bueno M, Marcos A; AVENA Study Group. Inflammatory proteins are related to total and abdominal adiposity in a healthy adolescent population: the AVENA Study. Am J Clin Nutr. 2006 Sep;84(3):505-12. doi: 10.1093/ajcn/84.3.505. PMID 16960163
- [Result] Adams MA, Roughley PJ. What is intervertebral disc degeneration, and what causes it? Spine (Phila Pa 1976). 2006 Aug 15;31(18):2151-61. doi: 10.1097/01.brs.0000231761.73859.2c. PMID 16915105